CLINICAL TRIAL: NCT03420339
Title: The Effects of Stimulant Medication on Disruptive Behavior, Choice, and Preference in Children and Adolescents Exhibiting Disruptive Behavior
Brief Title: Stimulant Effects on Disruptive Behavior
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Matthew J O'Brien, PhD, BCBA-D (Other)
Responsible Party: Sponsor-Investigator, Matthew J O'Brien, PhD, BCBA-D, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201709737
Record Dates: First submitted 2018-01-22; First posted 2018-02-05 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Attention Deficit Hyperactivity Disorder; Problem Behavior
Keywords: stimulant medication; behavioral function; preferences; delay discounting
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Problem Behavior | interventions — Central Nervous System Stimulants; Adderall; Methylphenidate; Dexmethylphenidate Hydrochloride; Lisdexamfetamine Dimesylate

STUDY DESIGN:
Intervention Model Description: In this study all participants will participate in behavioral assessments (i.e., preference assessments, functional analysis, choice assessments) while taking a stimulant medication and without taking a stimulant medication. All participants will experience the same protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects on stimulant medication (Experimental): All participants: Children and adolescents diagnosed with AD/HD, displaying disruptive behavior, and taking stimulant medication.
  Interventions: Drug: Stimulant

INTERVENTIONS:
Drug: Stimulant — The stimulants used must meet FDA dosage guidelines for age.
  Other Names: Adderall; Concerta; Aptensio; Daytrana; Metadate; Quillivant; Ritalin; Focalin; Vyvanse

SUMMARY:
The goal of this study is to determine the effects of stimulant medication on disruptive behavior, function, preference and choice; however, it is primarily methodological and will add to current research by establishing an effective evaluation of the impact of stimulant medication on these behaviors. Three behavior assessments for children and adolescents diagnosed with AD/HD who exhibit disruptive behavior will be conducted:

1. Preference assessments will be conducted to determine whether preference for social and nonsocial items and activities differs under medication and non-medication conditions.
2. Functional analyses will be conducted to determine whether stimulant medication has an effect on the frequency and function or purpose of disruptive behavior.
3. Choice assessments will be conducted to evaluate the impact of stimulant medication on impulse control/delay discounting.

This study will be conducted in three phases. For each of the 5 to 10 participants there will be 8 total visits. The first 4 visits will entail a preference assessment, followed by a functional analysis. On visits 1 and 3, the participant will be asked to take his/her stimulant medication as is typically done; however, on visits 2 and 4, the participant will be asked to refrain from taking the medication.

For visits 5-8, participants will continue to participate in preference assessments, but will also be presented with a choice arrangement with work and play. In the choice arrangement, participants will be given four work cards and four play cards that they can organize in any order. Work cards will be associated with a brief academic task and play cards will be associated with a brief play period using high-preferred toys/activities. On visits 5 and 7 the participant will be asked to take his or her stimulant medication as usual, while on visits 6 and 8 the participant will be asked to refrain from taking his or her medication.

DETAILED DESCRIPTION:
This study includes the consent, a pre-visit interview, and two assessment phases occurring at weekly visits. Phase I includes four visits, each lasting approximately 2 hours. Phase II includes four visits, each lasting approximately 1 hour. The following are the description of the consent, pre-visit, and Phases I and II:

Consenting:

A research team member will review eligibility criteria and study procedures with a prospective subject prior to requesting consent. Following consent, an interview will occur by phone or in person. If the caregiver desires, the interview may take place on the same visit as the consent (but following obtaining consent). In relation to the medication, withholding the medication will not occur until the second assessment visit (following the initial review and consent visit and also the interview).

Pre-Visit Interview:

If the interview is not conducted at the time of consent, it will be conducted either (a) at the first assessment visit, (b) by phone prior to the first visit or (c) in person prior to the first visit. The interview is standardized and gathers information on the subject's demographics, diagnosis/es, medications and stimulant medication history, disruptive behaviors and contexts, preferred items/activities, and common demands.

Phase I (visits 1, 2, 3,& 4):

Phase I of the study includes four visits total. Each visit will be conducted in the same manner and include three stages: (1) a free operant preference assessment, (2) a multiple stimulus without replacement preference assessment, and (3) three sessions of each test condition in a functional analysis. On visits 1 and 3 the subject will take his or her stimulant medication as expected before beginning the assessment procedures. Medications expected to have a delayed onset of action (e.g., Daytrana patch) will require the subject to take the medication greater than 60 minutes before the start of the assessments. On visits 2 and 4, the subject will withhold medication for the period he or she is completing the three stages. All data collection will be done using DataPal computer scoring software in the observation area of the therapy room. Each of these assessments is described next:

Stage 1: Free Operant Preference Assessment Upon arrival, the subject will enter the therapy room with a research team member, referred to as "researcher" henceforth. The therapy room will have no more than 10 items/activities, including up to 6 items/activities identified by the caregiver as "preferred", up to 2 items/activities selected by the researcher as potentially preferred, and up to 2 items/activities identified by the caregivers as neutral or "non preferred". The researcher will inform the subject that he or she may play with any of the items/activities within the therapy room. The researcher will make available his or her attention for the entirety of this portion of the assessment. No demands will be given to the subject and no consequences will be given for disruptive behavior. Data will be collected on the duration of item/activity engagement by the subject for each item/activity in the therapy room. This assessment will last 10 minutes. Items/activities with the greatest duration of engagement will be considered the highest preferred.

Stage 2: Multiple Stimulus Without Replacement within a Concurrent Operants Design Following the free operant preference assessment, 6 items/activities will be selected for another preference assessment. These items/activities will be available with and without attention. This preference assessment will be conducted in the same therapy room by the same researcher as the previous preference assessment. The assessment will begin by asking the subject to choose his or her most preferred item/activity to play with and with or without attention. The subject will be allowed 2 minutes with the item/activity and then it will be removed from the array. The subject will choose the next preferred item/activity with or without attention for another 2 minutes before removing that item/activity. This will continue until all items/activities have been selected (approximately 15 minutes). Data will be collected on the order of selection, attention or no attention, and engagement during the 2 minutes of access to each respective item/activity.

Stage 3: Functional Analysis of Problem Behavior

Following the preference assessments in Stages 1 and 2, a functional analysis of problem behavior will be conducted to determine the function(s) of the subject's problem behaviors. Disruptive behaviors will be deemed "target behaviors" for the functional analysis. All sessions of the functional analysis will be conducted by the researcher in the same therapy room as the previous two phases. Each session will last 5 minutes total, with 3 sessions for each test condition and 3 free play sessions. This results in a total of 12, 5-minute sessions, which may last between 75 to 90 minutes total. The order of conditions will be randomized for each round (i.e., one test of each condition and a free play session), with a newly randomized order for each round. The conditions include Escape, Tangible, Attention, and Free Play and are described below:

Free Play:

This condition serves as a control condition. Toys and activities will be available, as well as the researcher's attention. No work materials will be present. The researcher will begin the session by informing the subject that he/she may play with any toys/activities in the therapy room and that attention is available (e.g., "John, you can play with any of the toys in the room. I'll play with you if you like."). If a target behavior occurs (as well as any other "problem" behavior), the researcher will continue with attention and avoid commenting on the behavior.

Escape:

In this condition the subject will asked to complete demands. The demands will be (a) within the subject's skill range and (b) known to be aversive. This could be an academic task or a domestic task. The researcher will begin the session by presenting the demand to the subject using clear instructions (e.g., "John, it is time to do some math problems."). The researcher will provide praise as he/she is actively working. Attention will never be diverted. Tasks will continue to be presented unless a target problem behavior is observed. If a target behavior is emitted the researcher will provide a 30-second break from the work task. Once the 30-second break has ended the researcher will return to work using a prompt similar to that when the session started. For any subsequent occurrence of the target behavior there will be another break for 30 seconds. All non-target problem behaviors are ignored.

Tangible:

In this condition an item/activity identified as "high-preferred" and an item/activity identified as "low preferred" will be used. Just prior to the start of this condition, the subject is allowed access to the high-preferred item/activity. Once the session begins, the high-preferred item/activity will be restricted by the researcher and the low-preferred item/activity will be presented for play. Attention is not restricted during this condition. If the subject emits a target behavior the high-preferred item/activity is returned to the subject for 30 seconds and subsequently restricted again. If no target behavior occurs then the low-preferred item/activity will be the only play option for the entire five minutes.

Attention:

In this condition the subject has access to preferred items and activities and no demands are presented. At the beginning of the session the researcher will inform the subject that he or she should play with the toys available but that the attention will be unavailable. The researcher will leave the play area, go to the other side of the therapy room and begin reading a book or magazine. If a target behavior is emitted the researcher will approach the subject and provide a brief statement of disapproval and reiterate the expectation to behavior appropriately, followed by a return to ignoring the subject. All appropriate behavior, including requests for attention, will be ignored for the entirety of the session.

For the functional analysis, data will be collected and graphed on the frequency (rate per minute) of problem behavior. Visual inspection of graphs will determine differentiation across the four conditions (three test conditions and the freeplay/control condition) to identify the function(s) of the target behavior.

Phase II (visits 5, 6, 7, & 8):

Following completion of the first three stages (visits 1-4), four additional visits will be required (visits 5-8). These additional visits will consist of three stages: (1) free operant preference assessment; (2) multiple stimulus without replacement preference assessment in a concurrent operants design; and (3) work-break schedule with choice. Stages 1 and 2 will be conducted the same as Phase I. On visits 5 and 7 the subject will take his or her stimulant medication as expected before beginning and on visits 6 and 8, the subject will be asked to withhold medication for the period he or she is completing the three stages. All data collection will be done using DataPal computer scoring software that is installed on computers in the observation area of the therapy room.

Stage 1: Free Operant Preference Assessment This assessment will be conducted just as described for Phase I of the study.

Stage 2: Multiple Stimulus Preference Assessment within a Concurrent Operants Design This assessment will be conducted just as described for Phase I of the study.

Stage 3: Work-Play Schedule with Choice The purpose of this assessment is to evaluate delayed discounting and impulse control in choice making. In this stage, 8 picture cards and a schedule board (a plastic board with 8 Velcro placeholders for the picture cards) will be presented to the subject. Four of the picture cards will show a picture of a child working and the text "work". Four picture cards will depict a child playing and the text "play". Each "work" card will represent an academic work task. The worksheet(s) will take an estimated 5 minutes to complete Each "play" card will represent 3 minutes of play time with the high-preferred item/activity identified through the preference assessments in Stages 1 and 2. Attention will not be available during work or play; however, the subject may request help with the work if needed. Completion of the schedule will take approximately 32 minutes.

At the outset, the subject will be asked to organize the schedule in any sequence desired. There are many sequences the subject could choose (e.g., work(w)-play(p)-w-p-w-p-w-p; wwwwpppp, wwppwwpp, ppppwwww) and there will be no restriction on the sequence as long as all of the work and play cards are used in the sequence. Once the schedule is set by the subject the researcher will ask the subject to respond "final".

Following the sequencing of the schedule, the researcher direct and remind the subject of all transitions from one activity to the next. Each completed activity will result in the removal of the picture card from the schedule until all picture cards have been removed. The researcher will check the worksheets to ensure completion and will require the subject to complete any unfinished work items and redo incorrect work items until he or she has achieved 80% accuracy or better. Problem behavior will be placed on extinction (i.e., it will be ignored by the researcher and there will be no programmed consequences).. Data will be collected on the sequence chosen, compliance, on-task/off-task behavior, and problem behavior.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be a child or adolescent between the ages of 4 years, 0 months, and 13 years, 0 months (participants must not be older than 12 years, 11 months).
2. Participant must have a valid diagnosis of attention deficit/hyperactivity disorder (AD/HD). No specification of type (e.g., predominately inattentive type, predominately hyperactive-impulsive type, or combined type) will be necessary.
3. Participant must exhibit disruptive behavior, defined as one or more of the following:

   1. physical or verbal aggression towards others: Hitting, kicking, biting, scratching, choking, spitting at, or throwing items at another person, and/or making insults, threats, or swearing at another person.
   2. self-injury: Hitting self, biting self, banging head on an object/hard surface, pinching self, or scratching self with visual skin damage.
   3. destruction: Damaging (or attempts to damage) personal or public property (e.g., breaking an object into two or more pieces, using an object to break other objects, ripping objects or parts of objects from walls, floors, or furniture, and denting cars, objects, or walls.)
   4. noncompliance:Regular occurrence of verbal refusal (e.g., saying "no", "I don't want to", "I won't do it" or "not now") to any academic or non-academic request, and/or any response that does not match the delivered instruction within 30 seconds from the time the instruction was delivered.
   5. tantrum:Crying (i.e., any vocalizations [sounds or words] accompanied by facial contraction with and without tears for any period of time) and/or screaming (occurrence of vocalizations above normal conversational volume for any period of time), with or without body flailing.
   6. an active diagnosis of disruptive behavior disorder or oppositional defiant disorder.
4. Participant must already be prescribed a stimulant medication for the treatment of AD/HD symptoms and at an approved dose for age.

Exclusion Criteria:

1. a diagnosis of autism, conduct disorder, or intellectual disability in the moderate, severe or profound range.
2. prescribed or taking a stimulant dosage outside of recommended therapeutic range.

Ages: 48 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Behavioral Function | Weekly (at each visit): week 1, week 2, week 3, week 4; Change in behavioral function will be compared using data from weeks one and three (on medication) versus weeks two and four (off medication).
  Data will be collected and graphed on the frequency (rate per minute) of problem behavior. Visual inspection of graphs will determine differentiation across the four conditions (three test conditions and the freeplay/control condition) to identify the function(s) of the target behavior. Changes in behavioral function will be determined by comparing data week to week for the first four weeks. Behavioral function while on medication, which will occur at week one and week three will be compared to behavioral function at week two and week four. Differences between weeks one and three and weeks two and four will be considered as change in behavioral function.
Change in Item Preference | Weekly (at each visit): week 1, week 2, week 3, week 4, week 5, week 6, week, 7, week 8; we will compare data from weeks 1, 3, 5, and 7 (on medication) versus weeks 2, 4, 6, and 8 (off medication)
  Data on change in item preference will be collected week to week for all eight weeks. We will determine preference for an item/activity based upon the duration of time engaged with an item in the therapy room during the free operant preference assessment. Data will be compared week to week, with a focus on changes from weeks one, three, five, and seven (on medication) to weeks two, four, six, and eight (off medication). Differences in item engagement will indicate difference in item preference.
Change in Preference for Social and Non-Social Activities | Weekly (at each visit): week 1, week 2, week 3, week 4, week 5, week 6, week, 7, week 8; Changes in preference will be determined weekly, with a focus on differences between time points on medication and weeks off of medication.
  Data will be collected on the percentage of trials an activity is selected and whether it was selected with attention or without attention for each item/activity in the therapy room of the multiple stimulus without replacement assessment. Preference for social versus non-social activities will be determined by the participant's selection during the multiple stimulus without replacement assessment. The change in preference for activities with attention and activities without attention will be determined by comparing data weekly, with a focus on differences between data in weeks 1, 3, 5, and 7 (on medication) versus weeks 2, 4, 6, and 8 (off medication).
Changes in Impulsivity in Choice-Making | Weekly (at each visit): week 5, week 6, week 7, week 8
  Data will be collected on the sequence chosen by the subject and scored based upon the degree to which work sessions were placed up front and play activities were placed at the end. Choices whereby play activities are front loaded (i.e., more play activities earlier in the schedule) will be scored as more impulsive on a point system and choices whereby work activities are front loaded (i.e., more work activities earlier in the schedule) will be scored as less impulsive. Differences in impulsivity will be determined on a week to week basis, with a focus on differences between weeks on medication (weeks 5 and 7) and weeks off of medication (weeks 6 and 8).

SECONDARY OUTCOMES:
Rate of Problem Behavior | Weekly (at each visit): week 1, week 2, week 3, week 4, week 5, week 6, week, 7, week 8
  Data will be collected in all assessment sessions on the rate of problem behavior and compared for sessions on medication and sessions off medication.
Item Engagement | Weekly (at each visit): week 1, week 2, week 3, week 4, week 5, week 6, week, 7, week 8
  Data will be collected in all assessment sessions involving play with items/activities on item engagement and compared for sessions on medication and sessions off medication.
Compliance | Weekly (at each visit): week 1, week 2, week 3, week 4, week 5, week 6, week, 7, week 8
  Data will be collected on compliance to demands for all sessions involving work. Data will be compared for sessions sessions on medication and sessions off medication.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J O'Brien, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No